CLINICAL TRIAL: NCT07055217
Title: Effect of Mindfulness-based Neurofeedback for Adolescents With Elevated Repetitive Negative Thinking
Acronym: CHARMS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Anne Eden Evins, Cox Family Professor of Psychiatry, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2025P001338; R61MH139856 (NIH)
Record Dates: First submitted 2025-06-10; First posted 2025-07-08 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-11

CONDITIONS: Repetitive Negative Thinking; Neurofeedback
Keywords: Adolescents at risk for serious mental illness; Mindfulness; Real-time fMRI; Neurofeedback; DMN Connectivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy Control (HC) (No Intervention): Healthy control participants will complete a brief resting state MRI scan at Visit 2 to assess default mode network connectivity. They will receive no intervention or comparator.
- Mindfulness-based neurofeedback (mbNF) (Experimental): Participants will:
  * Complete a brief resting state MRI scan at Visit 2 to assess default mode network connectivity
  * Receive a 45-minute mindfulness training
  * Receive two 15-minute sessions of mindfulness-based neurofeedback
  Interventions: Behavioral: Mindfulness Training; Behavioral: Mindfulness-based Neurofeedback (Real mbNF)
- Sham mindfulness-based neurofeedback (Sham mbNF) (Sham Comparator): Participants will: - Complete a brief resting state MRI scan at Visit 2 to assess default mode network connectivity -Receive a 45-minute mindfulness training -Receive two 15-minute sessions of sham mindfulness-based neurofeedback
  Interventions: Behavioral: Mindfulness Training; Behavioral: Sham mindfulness-based neurofeedback (Sham mbNF)

INTERVENTIONS:
Behavioral: Mindfulness Training — A single 45-minute mindfulness training will be provided to all at-risk participants at visit 2. Clinically trained study staff will conduct the training with the aim of teaching "mental noting," a core mindfulness technique to be practiced and employed during neurofeedback. Mental noting is a major component of Vipassana (insight mindfulness meditation); its key principles include: "concentration", "observing sensory experience,'' "not 'efforting'", and "contentment".Specifically, participants will be taught to mentally label/note whatever sensation is most prominent in their sensory experience from moment to moment (e.g., seeing, hearing, feeling, thinking). Training will be personalized to identify scenarios in which mental noting can be applied in the context of each person's daily life, explaining the goal of using these strategies to manage distress in daily life.
  Arms: Mindfulness-based neurofeedback (mbNF); Sham mindfulness-based neurofeedback (Sham mbNF)
Behavioral: Mindfulness-based Neurofeedback (Real mbNF) — Before the MRI scan, participants will practice mental noting by verbalizing their mental label, with the study clinician providing feedback. Participants will then complete a silent practice of mental noting while viewing simulated neurofeedback. All participants will be trained until they feel competent to use mental noting in the scanner. Study clinicians will show 85% fidelity on the mindfulness training assessment before working with participants and sessions will be recorded and 10% of sessions will be assessed quarterly for fidelity. During active mbNF (6 runs, 2.5 mins each), participants will use mental noting with the aim of controlling the visual feedback; specifically, they will attempt to move the position of the white dot toward the (upper) red circle and away from the (lower) blue circle.
  Arms: Mindfulness-based neurofeedback (mbNF)
Behavioral: Sham mindfulness-based neurofeedback (Sham mbNF) — During sham mbNF condition, participants will undergo similar MRI scan procedures. The primary difference in scan procedures is that rather than receiving mbNF, participants will view a visual display (i.e., white dot, red and blue circles) extracted from a previously acquired mbNF session. Thus, the visual display will be independent from brain activity in the sham condition and will simply mirror the stimuli observed by those in the mbNF group. This ensures that participants across groups are viewing equivalent stimuli for the same amount of overall time.
  Arms: Sham mindfulness-based neurofeedback (Sham mbNF)

SUMMARY:
This study will test the hypotheses that adolescent with repetitive negative thinking who at at-risk for serious mental illness will show greater default mode network (DMN) connectivity than healthy controls, at-risk adolescents will show greater changes in DMN connectivity than healthy controls, and that a longer session of mindfulness based neurofeedback will lead to greater reduction in DMN connectivity. To do so, 50 adolescents with elevated repetitive negative thinking and 50 matched healthy control participants will be enrolled into a double-blind randomized clinical trial of a session of mindfulness training with either active mindfulness-basde neurofeedback or sham mindfulness-based neurofeedback.

DETAILED DESCRIPTION:
A sample of 50 at-risk adolescents with elevated repetitive negative thinking and 50 matched healthy control participants, ages 13-21, will be enrolled into this double blind, randomized clinical trial. Healthy control participants will be matched for age and sex. All participants will complete a baseline clinical assessment and return within two weeks for a brief resting state MRI scan to assess default mode connectivity (DMN). At Visit 2, at-risk adolescents will then receive a 45-minute mindfulness training by clinically trained staff. After the mindfulness training, participants will be randomized in a 1:1 ratio to receive either active or sham neurofeedback. Participants and staff will remain blind to assignment. Participants will have fMRI scans for resting state functional connectivity before and after mindfulness practice. Participants will complete two doses (15 minutes per dose) of real or sham mbNF in the scanner. At-risk adolescents will also complete a follow-up clinical assessment at 4-weeks post-scan (Visit 3) and complete daily surveys for approximately four weeks from Visit 2 to Visit 3.

ELIGIBILITY:
Inclusion Criteria:

* Ages 13-21, inclusive
* If <18 years old: Competent and willing to provide written informed assent AND have a parent/legal guardian who is competent and willing to provide written informed consent
* If age ≥18 years: Competent and willing to provide written informed consent
* Tanner puberty stage ≥3 (to minimize neuroendocrine variability)
* Able to understand study procedures, read, and write in English
* Access to a mobile device to complete daily surveys

Additional Inclusion Criteria for At-Risk Adolescents - Recurrent negative thinking, defined as PTQ/PTQ-C total score >30 with at least two items rated as 3 (Often) or 4 (Almost Always)

Additional Inclusion Criteria for Healthy Controls

-PTQ/PTQ-C total score <15, with zero items rated as 3 (Often) or 4 (Always)

Exclusion Criteria:

* Any of the following lifetime mental health disorders by DSM-V criteria: psychotic disorders, bipolar disorder, moderate, severe or recurrent major depressive disorder, conduct disorder, developmental disorder (e.g., autism), post-traumatic stress disorder, or obsessive compulsive disorder
* Severe lifetime substance use disorder
* Unstable medical or neurologic condition as determined by study staff, history of epilepsy or seizure disorder, head injury, loss of consciousness >5 minutes by participant self-report
* MRI contraindications (i.e. presence of ferromagnetic implants, cardiac pacemaker or pacemaker wires, metallic particles in the body, vascular clips in the head or previous neurosurgery, prosthetic heart valves, magnetic dental implants claustrophobia).
* Visual, auditory, or cognitive impairment (IQ<80 based on the Wechsler Abbreviated Intelligence Scale (WASI)) that may make it difficult to participate.
* Any condition or situation that would, in the investigator's opinion, make it unlikely that the participant could adhere safely to the study protocol.
* Pregnancy: a negative pregnancy test is required at the time of enrollment for any individuals of childbearing potential
* Individuals who are under the legal protection of the government or state (Wards of the State)

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Resting State Default Mode Network (DMN) Functional Connectivity | Baseline
  We will test whether at-risk adolescents have higher default mode network (DMN) functional connectivity (i.e., hyperconnectivity) compared to healthy control participants. A matched-sample t-test will examine baseline functional connectivity between two canonical DMN nodes (personalized medial prefrontal cortex and posterior cingulate cortex).
Change in Within-Person Default Mode Network (DMN) Functional Connectivity | Pre-mbNF, Post-mbNF (30 minutes after pre-mbNF)
  A repeated measures ANCOVA will test interaction between within-participant change (2-level factor: pre- vs. post-mbNF) and between participant contrast (2-level: real- vs. sham-mbNF) in functional connectivity between two canonical DMN nodes (personalized medial prefrontal cortex and posterior cingulate cortex) as the dependent measure.
Time Effect on Within-DMN Connectivity | Pre-mbNF, First post-mbNF (15 minutes after pre-mbNF), Second post-mbNF (30 minutes after pre-mbNF)
  A repeated-measures ANCOVA will be used to test potential effect of time (three within-participant levels: pre-mbNF, first post-mbNF (15 minutes), second post-mbNF (30 minutes)) on functional connectivity between two canonical DMN nodes (personalized medial prefrontal cortex and posterior cingulate cortex).

CONTACTS AND LOCATIONS:
Overall Officials: A. Eden Evins, MD, MPH, Principal Investigator — Massachusetts General Hospital; Susan Whitfield-Gabrieli, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Center for Addiction Medicine, 101 Merrimac Street, Suite 320, Boston, MA 02114, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Data from this study will be submitted to the National Institute of Mental Health Data Archive (NDA). NDA is a large database where de-identified study data from many NIH-funded studies are stored and managed. The final dataset to be shared will include demographic, clinical (diagnostic interviews, questionnaires), and neuroimaging (MRI and fMRI) data collected from at-risk adolescents and healthy controls. Sufficient data from this project to validate and replicate findings described in the aims will be shared. The study protocol will be published as a methods/protocol paper. We will also publish and maintain detailed neurofeedback experiment data (including stimuli, experiment scripts, and analysis scripts) on GitHub.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Scientific data will be available one year after the grant end date specified on the first Notice of Award. Scientific data included in published manuscripts will be available at the time of publication if the publication occurs before the end of the grant period. NDA will make decisions about how long to preserve the data.
Access Criteria: To request access of the data, researchers will use the standard processes at NDA, and the NDA Data Access Committee will decide which requests to grant. The standard NDA data access process allows access for one year and is renewable.